CLINICAL TRIAL: NCT06659133
Title: In Women Undergoıng Paddle Endometrıal Bıopsy Applıed Musıc Recıtal Effect On Paın And Anxıety
Brief Title: Effect of Music On Pain and Anxiety Paddle Edometrial Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Didem Kucukkelepce, Phd, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: lokmanhekim universty
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Gynecologic Nursing
Keywords: pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study was conducted as a randomized controlled trial to investigate the effect of music recital on pain and anxiety in women undergoing pipelined endometrial biopsy.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): control group received routine care during pipelined endometrial biopsy.
- Music (Experimental): The experimental group listened to acemashiran maqam music during pipelined endometrial biopsy.
  Interventions: Other: Music intervention

INTERVENTIONS:
Other: Music intervention — The women participating in the study were divided into control and experimental groups.
  The control group included women who underwent pipelle endometrial biopsy with routine care, and the experimental group included women who underwent pipelle endometrial biopsy accompanied by music. Pipelle endometrial biopsy was performed by the same physician working in the Department of Obstetrics and Gynecology at the hospital. Patients in both groups were interviewed 10 minutes before the endometrial biopsy procedure and the Personal Information Form and State and Trait Anxiety Scale were applied. The application of the GKO was explained to the patients before the pipelle endometrial biopsy procedure. Before the pipelle endometrial biopsy, all patients were routinely given local anesthesia with 8 cc of 2% lidocaine solution and waited for 5 minutes after the application of local anesthesia.
  During the pipelle endometrial biopsy, the experimental group was given a music recital from an mp3 play
  Arms: Music

SUMMARY:
This study was conducted as a randomized controlled trial to investigate the effect of music recital on pain and anxiety in women undergoing pipelined endometrial biopsy.

DETAILED DESCRIPTION:
This study was conducted as a randomized controlled trial to investigate the effect of music recital on pain and anxiety in women undergoing pipelined endometrial biopsy. The data were collected in the intervention room of the mixed service of a state hospital in Ankara between December 2023 and April 2024. Power analysis was performed with the G*Power 3.1 program to determine the number of people to be included in the study. The study was conducted with a total of 64 women, 32 in the control group and 32 in the experimental group. The data were collected using the Personal Information Form, "Visual Comparison Scale" to assess the severity of pain, and "State and Trait Anxiety Scale" to determine the level of anxiety. The experimental group listened to acemashiran maqam music, while the control group received routine care. There was no significant difference between the control and experimental groups in the distribution of socio-demographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over who underwent endometrial biopsy for the first time

Exclusion Criteria:

Those who did not fill out the consent form, Those who were illiterate, Those who were receiving inpatient treatment during the study, Those with psychiatric illness (dementia, psychosis, etc.), Those who were on regular medication (such as analgesics, anxiolytics or sedatives), Those who had communication problems (vision, hearing and perception problems), Women who were in pain before the procedure were not included.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 64 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
anxiety | 30 min
  State and Trait Anxiety Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Didem Simsek Kucukkelepce, Adıyaman, Turkey (Türkiye)